CLINICAL TRIAL: NCT06663969
Title: Evaluating Modulation Effects of Temporal Interference Using SEEG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Liankun_Ren, Professor, Xuanwu Hospital, Beijing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2024-258-002
Record Dates: First submitted 2024-10-26; First posted 2024-10-29 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Deep Brain Stimulation; Drug Resistant Epilepsy
Keywords: Temporal Interference; Stereoelectroencephalography; Drug Resistant Epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Temporal Interference (Experimental): The investigators performed temporal interference (TI) stimulation to patients with drug-resistant epilepsy undergoing SEEG monitoring. They observed electrophysiological activity and clinical manifestations before, during, and after stimulation to investigate the electrophysiological mechanisms of TI.
  Interventions: Other: Temporal Interference

INTERVENTIONS:
Other: Temporal Interference — Researchers applied temporal interference (TI) stimulation to the deep brain nuclei of patients who had undergone SEEG monitoring, recording changes in electrical activity detected by SEEG.

SUMMARY:
This single-center prospective study aims to investigate the electrophysiological mechanisms of temporal interference (TI) in humans by analyzing clinical, imaging, and electrophysiological data from patients aged 14-60 with drug-resistant epilepsy.

DETAILED DESCRIPTION:
Temporal Interference (TI) technology is a novel non-invasive method for deep brain stimulation (DBS). By generating an overlapping electric field from safe currents, TI creates focused stimulation in targeted deep brain areas. This approach allows for the exploration of deep brain nuclei functions and has the potential to serve as a non-invasive alternative to traditional invasive DBS for clinical treatments.

Stereoelectroencephalography (SEEG) is a method for recording electrical activity from deep brain structures using implanted depth electrodes to provide a three-dimensional view of neuronal activity.

This study aims to investigate the electrophysiological mechanisms of temporal interference (TI) deep brain stimulation by including patients aged 14-60 with implanted intracranial electrodes. During and after TI stimulation, electrophysiological and clinical data will be recorded. Clinical, imaging, and electrophysiological data will be analyzed and processed to advance understanding of TI's effects in deep brain stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of drug-resistant epilepsy;
* No severe systemic diseases;
* Implantation of stereotactic electrodes;
* Agreement to participate in this study and signs the informed consent form.

Exclusion Criteria:

* Hematoma at the scalp electrode site or fluid accumulation under the electrode after intracranial electrode placement.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Electrophysiological changes | During the trial(up to 3 hours for each subject)
  Electrophysiological waveform changes recorded by stereoelectroencephalography (SEEG) before, during, and after TI stimulation.

SECONDARY OUTCOMES:
Patient's subjective feelings and symptoms | During the trial(up to 3 hours for each subject)
  Researchers categorized patients' clinical responses as normal, mild, moderate, or severe based on their subjective clinical response.

CONTACTS AND LOCATIONS:
Overall Officials: Liankun Ren, MD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital,Capital Medical University, Beijing, Beijing Municipality, China